CLINICAL TRIAL: NCT05138601
Title: Remote Monitoring and Virtual Collaborative Care For Hypertension Control to Prevent Cognitive Decline Phase II
Acronym: vCCC 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Utah (Other); University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00147392
Record Dates: First submitted 2021-09-22; First posted 2021-12-01 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care with Education (No Intervention): The participant will be provided with educational material and a home BP monitor. Control participants will continue to see their physicians for their usual care for BP management (their BP data will not be reviewed by pharmacists and the patients will not have support from vCCC pharmacists)
- Virtual Collaborative Care Clinic (Experimental): Participants will partake in the virtual collaborative care clinic
  Interventions: Other: Virtual Collaborative Care Clinic

INTERVENTIONS:
Other: Virtual Collaborative Care Clinic — Trained clinical pharmacists will monitor BP, prescribe and adjust medications and monitor for side effects of medications under the license of, and in communication with, the patient's physician.
  Arms: Virtual Collaborative Care Clinic

SUMMARY:
This is a randomized, controlled, pragmatic trial designed as a "type I hybrid effectiveness-implementation trial" that tests a hypertension program integrating a virtual Collaborative Care Clinic (vCCC), home blood pressure monitoring, and telehealth for lowering blood pressure (BP) in two health systems.

DETAILED DESCRIPTION:
This study tests a hypertension program integrating a virtual Collaborative Care Clinic (vCCC), home blood pressure monitoring, and telehealth for lowering blood pressure (BP) in two health systems (University of Kansas Health System [UKHS] and the University of Utah Health [UUtah]). The vCCC is staffed by clinical pharmacists who remotely monitor home BP and use telehealth to work with patients to lower systolic blood pressure (SBP) to <130 mmHg, as recommended by the current American College of Cardiology/American Heart Association (ACC/AHA) guidelines. Eligible patients with uncontrolled hypertension (HTN) are identified automatically through the electronic health record (EHR) during visits to their Primary Care Provider (PCP) and referred for enrollment into the vCCC.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* Active patient in participating primary care clinic
* Access to compatible "smartphone" or device (i.e., Android, Kindle or Apple with internet connectivity or mobile network)
* Elevated BP as defined by
* SBP >140 at current visit AND documented history of hypertension OR SBP > 140 at current visit and at another visit in last 18 months OR SBP >160 at current visit
* Sufficiently fluent in English to participate in study procedures
* Adequate hearing to complete study procedures
* Able to give their own signed consent
* Health insurance coverage by Medicare

Exclusion Criteria:

* Clinically significant illness that may affect safety or completion per their treating PCP or study physician
* Needing interpreter for clinic visits (through Electronic Health Record)
* Currently in hospice care
* Currently receiving chemotherapy
* Unable to take accurate BP measurement, either due to inability to follow protocol to check BP or due to medical conditions such as lymphedema or dialysis access on both arms.
* Currently participating in another intervention trial
* End stage kidney disease on dialysis
* Diagnosis of dementia (i.e., dementia, Alzheimer's disease, vascular dementia, dementia with Lewy bodies, frontotemporal dementia)
* Chronic active disease with expected life expectancy < 2 years as determined by the study team

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure (SBP) Control At 24 Months | 24 months.
  Our primary outcome is achieving SBP control (<130 mmHg). Blood pressure measures will be collected in a dashboard system and will be integrated into the common data model table for final analysis. Investigators will utilize the Benjamini-Hochberg approach to control for multiple testing in our primary outcome.

SECONDARY OUTCOMES:
Cognitive Measures | 0 months, 12 months, and 24 months
  Investigators will use composite z score obtained by averaging standardized z scores of individual NP test scores and use z scores of individual tests to determine changes in a single test that may be obscured with the measurement of a global score. The tests are Montreal Cognitive Assessment (MoCA) Blind, Rey Auditory Verbal Learning Test (RAVLT), Number Span Forwards and Backwards (NSFB), Oral Trail Making Test (OTMT), Category Fluency, Verbal Fluency, Rey Auditory Verbal Naming Test Delayed Recall and Recognition, and Verbal Naming Test (VNT). MoCA Blind has 22 possible points, with19 or above normal. NSFB gives 2 scores, total number of correct trials and longest sequence repeated correctly with higher score indicating better working memory. The category fluency has 2 possible scores with a higher number of unique names indicating a better semantic memory. For the Verbal Fluency test the score reflects the number of unique responses with a higher score indicating better memory
Major Adverse Cardiovascular Events (MACE) | 24 months
  Data from the electronic health record (EHR) will be extracted. MACE will be identified by will be identified by International Statistical Classification of Diseases and Related Health Problems (ICD) and Current Procedural Terminology (CPT) codes for hospitalization due to myocardial infarction (MI), nonfatal stroke, coronary revascularization, and heart failure, which will be identified by combining observations from EHR
Atherosclerotic Cardiovascular Disease Risk (ASCVD) | 24 months
  Data from the EHR will be extracted. (ASCVD) score will be estimated by age, sex, race, BP, total cholesterol, HDL cholesterol, history of diabetes, smoking status, HTN treatment, statin and aspirin therapy. ASCVD score is given as a percentage. A 0 to 4.9% risk is considered low risk, 5 to 7.4% is considered borderline, a 7.5 to 20% risk is considered intermediate, and a score above 20% is considered high.
Health Care Resource Utilization: Charges Per Patient | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include charges per patient (measured as total and average dollar amount of charges).
Mortality | 2 years
  All-cause mortality, as a composite endpoint, will be obtained from Common Data Model DEATH table and be ascertained by linked Medicare Beneficiary Summary File available from Centers for Medicare and Medicaid Services (CMS)
Systolic Blood Pressure (SBP) Control At 12 Months | 12 Months
  Our primary outcome is achieving SBP control (<130 mmHg). Blood pressure measures will be collected in a dashboard system and will be integrated into the common data model table for final analysis. Investigators will utilize the Benjamini-Hochberg approach to control for multiple testing in our primary outcome.
Health utilization outcome measurement: Carrier Claims | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include healthcare-facility-metrics, such as carrier (physician Part B) claims (measured as total and average counts of distinct claims)
Health utilization outcome measurement: facility claims | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include outpatient, inpatient, skilled nursing facility claims (measured as total and average counts of distinct claims).
Health utilization outcome measurement: coronary care claims | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include component-of-care metrics, such as coronary care claims (measured as total and average counts of distinct claims)
Health utilization outcome measurement: coronary care expenditures | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include component-of-care metrics, such as coronary care expenditures (measured as total and average dollar amount of charges) per patient
Health utilization outcome measurement: coronary care unit days | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include component-of-care metrics, such as coronary care unit days (measured as total length of stay in coronary care unit).
Health utilization outcome measurement: intensive care unit (ICU) days | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include component-of-care metrics, such as ICU days (measured as total length of ICU stay) per patient.
Health utilization outcome measurement: general drug claims | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include component-of-care metrics such as general drugs and/or IV therapy claims (measured as total and average counts of distinct claims) per patient.
Health utilization outcome measurement: durable medical equipment Medicare payments | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include component-of-care metrics such as durable medical equipment Medicare payments (measured as total and average dollar amount of charges) per patient.
Health utilization outcome measurement: imaging and laboratory events | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include component-of-care metrics such as imaging and laboratory events (measured as total and average counts of distinct claims suggesting imaging and laboratory events).
Health utilization outcome measurement: imaging and laboratory expenditures | 2 years
  Health utilization outcome measurement will be ascertained mainly by CMS claims data. The utilization outcome measurement will include component-of-care metrics such as imaging and laboratory expenditures (measured as total and average dollar amount of charges) per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Burns, MD, MS, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Health System, Kansas City, Kansas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No